CLINICAL TRIAL: NCT01868919
Title: Implementation Research of a Parenting Intervention to Improve Behaviour in Children in Primary Care
Brief Title: Triple P to Improve Behaviour in Children
Acronym: TriplePChile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TRIPLEP.PUC.CHILE
Record Dates: First submitted 2013-01-19; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Parenting; Child Behaviour; Mental Health Wellness 1; Family Research
Keywords: "Pilot Projects"[Mesh]; "Parenting"[Mesh]; "Child Behaviour"[Mesh]; "Mental Health"[Mesh]; "Family Practice"[Mesh]
MeSH Terms: interventions — (tris(diphenylphosphinomethyl)phenylborate)(p-tolylnitrido)iron(I)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive Parenting Program (Experimental): Level 3 or 4 of Triple P
  Interventions: Behavioral: Positive Parenting Program

INTERVENTIONS:
Behavioral: Positive Parenting Program — Level 3 or 4 of Triple P
  Other Names: Triple P

SUMMARY:
Joint research (quantitative and qualitative methodology) with quasi-experimental design, before-after without control group to evaluate the pilot implementation of Positive Parenting Program (Triple P) in the context of primary health care in Chile. The hypothesis is that the program is feasible and acceptable to the Chilean population.

DETAILED DESCRIPTION:
General Purpose:

● Evaluate the pilot implementation of the Triple P program in the context of primary health care in Chile.

Specific Objectives:

1. To assess the fidelity of implementation of the Triple P program
2. Analyze the perception of participants, providers and organization on determinants of program implementation.
3. Identify barriers and facilitators to plan future implementation of Triple P program in contexts similar to those in the study.
4. To estimate the magnitude of change in children's behavior, emotional difficulties and rearing practices of caregivers before and after participation.

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregivers of children from 2 to 10 years old attending primary care clinic
* Parents or caregivers must be worried about child behaviour or their parenting skills and be willing to get professional help

Exclusion Criteria:

* Children: Pervasive Developmental Disorder, severe intellectual disability or severe psychopathology
* Caregivers: illiteracy, decompensated severe psychopathology or current psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Assess implementability of the program in primary care in terms of feasibility, acceptability and level of participation | After one year of implementation
  Instrument: focus groups

SECONDARY OUTCOMES:
Percentage of change in intensity of behaviour in children | After one year of implementation
  Instrument: Eyberg Child Behaviour Inventory
Fidelity of program implementation | After one year of implementation
  Supervision meetings and video recordings

CONTACTS AND LOCATIONS:
Overall Officials: Gladys Moreno, Dra., Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- See also: Triple P Chilean website — http://www.triplep.cl
- See also: Triple P Official Website — http://www.triplep.net
- See also: Triple P Provider Network — http://www.triplep.org